CLINICAL TRIAL: NCT04411641
Title: A Phase 3, Randomized, Double-blind, Efficacy and Safety Study Comparing SAR442168 to Placebo in Participants With Nonrelapsing Secondary Progressive Multiple Sclerosis
Brief Title: Nonrelapsing Secondary Progressive Multiple Sclerosis (NRSPMS) Study of Bruton's Tyrosine Kinase (BTK) Inhibitor Tolebrutinib (SAR442168) (HERCULES)
Acronym: HERCULES
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: EFC16645; U1111-1246-7768 (Registry Identifier: ICTRP); 2020-000647-30 (EudraCT Number)
Record Dates: First submitted 2020-05-28; First posted 2020-06-02 (Actual); Results first posted 2025-06-18 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-06

CONDITIONS: Non-relapsing Secondary Progressive Multiple Sclerosis

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- SAR442168 (Experimental): 60 mg of oral SAR442168 once daily
  Interventions: Drug: Tolebrutinib
- Placebo (Placebo Comparator): Placebo tablet to match SAR442168 once daily
  Interventions: Drug: Placebo to match Tolebrutinib

INTERVENTIONS:
Drug: Tolebrutinib — Pharmaceutical form: Film-coated tablet Route of administration: Oral
  Other Names: SAR442168
  Arms: SAR442168
Drug: Placebo to match Tolebrutinib — Pharmaceutical form: Film-coated tablet Route of administration: Oral
  Arms: Placebo

SUMMARY:
Primary Objective:

To determine the efficacy of SAR442168 compared to placebo in delaying disability progression in NRSPMS

Secondary Objective:

To evaluate efficacy of SAR442168 compared to placebo on clinical endpoints, magnetic resonance imaging (MRI) lesions, cognitive performance, physical function, and quality of life To evaluate safety and tolerability of SAR442168 To evaluate population pharmacokinetics (PK) of SAR442168 and relevant metabolites in NRSPMS and its relationship to efficacy and safety To evaluate pharmacodynamics (PD) of SAR442168

DETAILED DESCRIPTION:
This was an event-driven (6-month CDP) trial with a variable treatment duration (end-of-study [EOS] duration: up to approximately 47months).

Participants with 6-month confirmed disability progression (CDP) had an option to receive tolebrutinib in the open-label (OL).

ELIGIBILITY:
Inclusion criteria :

* 18 to 60 years of age inclusive
* Diagnosis of nonrelapsing secondary progressive multiple sclerosis according to the 2017 McDonald criteria
* Expanded disability status scale (EDSS) between 3.0 to 6.5 points inclusive, at screening
* The participant must have documented evidence of disability progression observed during the 12 months before screening
* Absence of clinical relapses for at least 24 months
* Contraceptive use by men or women should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies
* A female participant is eligible to participate if she is not pregnant or breastfeeding, and at least one of the following conditions applies:
* Is not a WOCBP OR
* Is a WOCBP and agrees to use an acceptable contraceptive method

Exclusion criteria:

* The participant has conditions that would adversely affect study participation such as short life expectancy.
* Evidence of infection with human immuodeficiency virus (HIV), transplantation, progressive multifocal leukoencephalopathy (PML), active hepatitis B or C, active or latent tuberculosis or other active infections that would adversely affect study participation.
* Persistent chronic or active or recurring system infection, that may adversely affect participation or IMP administration in this study, as judged by the Investigator.
* History of malignancy within 5 years prior to screening.
* History of alcohol or drug abuse within 1 year prior to screening.
* Hospitalized for psychiatric disease within 2 years prior to screening.
* Clinically significant laboratory abnormalities (including evidence of liver injury) or electrocardiogram abnormalities at screening
* Bleeding disorder, known platelet dysfunctionat any time prior to the screening visit
* A platelet count <150 000/μL at the screening visit
* A history of significant bleeding event within 6 months prior to screening, according to the Investigator's judgment such as, but not limited to cerebral or gastrointestinal bleeding.
* Lymphocyte count below the lower limit of normal at screening.
* Recent live (attenuated) vaccine within 2 months before the first treatment visit.
* Recent major surgery (within 4 weeks of screening) or planned major surgery during the study.
* The participant has received medications/treatments for MS within a specified time frame.
* Receiving potent and moderate inducers or inhibitors of cytochrome P450 3A (CYP3A) or potent inhibitors of CYP2C8 hepatic enzymes.
* Receiving anticoagulant or antiplatelet therapy (such as aspirin>81mg/day, clopidogrel, warfarin).
* Contraindications to magnetic resonance imaging (MRI).

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1131 (Actual)
Dates: Start 2020-09-24 (Actual); Primary Completion 2024-08-29 (Actual); Study Completion 2024-08-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (306):
- United States (51):
  - University of Alabama MS Center-Site Number:8400013, Birmingham, Alabama
  - Center for Neurology and Spine-Site Number:8400089, Phoenix, Arizona
  - Arcadia Neurology Center-Site Number:8400070, Arcadia, California
  - UC San Diego ACTRI-Site Number:8400101, La Jolla, California
  - Collaborative Neuroscience Research-Site Number:8400045, Long Beach, California
  - Multiple Sclerosis Center-Site Number:8400143, Los Angeles, California
  - University of San Francisco, Sandler Neurosciences Center-Site Number:8400137, San Francisco, California
  - Harbor UCLA-Site Number:8400088, Torrance, California
  - Regina Berkovich, MD, PhD-Site Number:8400059, West Hollywood, California
  - Mountain Neurological Research Center, Inc.-Site Number:8400128, Basalt, Colorado
  - University of Colorado-Site Number:8400012, Denver, Colorado
  - Advanced Neurosciences Research-Site Number:8400025, Fort Collins, Colorado
  - South Florida Neurology Associates-Site Number:8400029, Boca Raton, Florida
  - Neurology Associates, PA-Site Number:8400004, Maitland, Florida
  - Aqualane Clinical Research-Site Number:8400027, Naples, Florida
  - Axiom Clinical Research of Florida-Site Number:8400001, Tampa, Florida
  - University of South Florida-Site Number:8400006, Tampa, Florida
  - Meridian Clinical Research-Site Number:8400003, Savannah, Georgia
  - Consultants In Neurology-Site Number:8400011, Northbrook, Illinois
  - University of Kansas Medical Center-Site Number:8400023, Kansas City, Kansas
  - CHI Saint Joseph Medical Group Neurology-Site Number:8400110, Lexington, Kentucky
  - Tufts Medical Center-Site Number:8400072, Boston, Massachusetts
  - University of Massachusetts-Site Number:8400014, Worcester, Massachusetts
  - Wayne State University-Site Number:8400046, Detroit, Michigan
  - The Memorial Hospital-Site Number:8400033, Owosso, Michigan
  - Minneapolis Clinic of Neurology-Site Number:8400051, Minneapolis, Minnesota
  - Mayo Clinic-Site Number:8400111, Rochester, Minnesota
  - Missouri Baptist Medical Center-Site Number:8400019, St Louis, Missouri
  - Lou Ruvo Center for Brain Health-Site Number:8400117, Las Vegas, Nevada
  - Holy Name Hospital-Site Number:8400104, Teaneck, New Jersey
  - University of New Mexico-Site Number:8400032, Albuquerque, New Mexico
  - Icahn School of Medicine at Mount Sinai (Department of Endoc-Site Number:8400038, New York, New York
  - Neurology Associates of Stony Brook-Site Number:8400042, Stony Brook, New York
  - Meridian Clinical Research, LLC-Site Number:8400005, Raleigh, North Carolina
  - Sanford Brain & Spine Center-Site Number:8400126, Fargo, North Dakota
  - University Hospitals CMC-Site Number:8400083, Cleveland, Ohio
  - Cleveland Clinic-Site Number:8400125, Cleveland, Ohio
  - Optimed Research, LTD-Site Number:8400147, Columbus, Ohio
  - Neurology Specialists-Site Number:8400002, Dayton, Ohio
  - Columbus Neuroscience-Site Number:8400010, Westerville, Ohio
  - Providence Multiple Sclerosis Center-Site Number:8400020, Portland, Oregon
  - Perelman Center for Advanced Medicine-Site Number:8400142, Philadelphia, Pennsylvania
  - Jefferson Neurology Associates-Site Number:8400016, Philadelphia, Pennsylvania
  - Premier Neurology-Site Number:8400069, Greer, South Carolina
  - Mountain View Clinical Research-Site Number:8400024, Greer, South Carolina
  - Neurology Clinic, PC-Site Number:8400087, Cordova, Tennessee
  - Advanced Neuroscience Center-Site Number:8400035, Franklin, Tennessee
  - Baylor College of Medicine-Site Number:8400136, Houston, Texas
  - Neurology Center of San Antonio-Site Number:8400036, San Antonio, Texas
  - University Of Vermont College Of Medicine-Site Number:8400130, Burlington, Vermont
  - Medical College of Wisconsin-Site Number:8400028, Milwaukee, Wisconsin
- Argentina (5):
  - Investigational Site Number :0320002, Capital Federal, Buenos Aires
  - Investigational Site Number :0320001, CABA, Buenos Aires F.D.
  - Investigational Site Number :0320007, Buenos Aires
  - Investigational Site Number :0320006, Córdoba
  - Investigational Site Number :0320005, San Miguel de Tucumán
- Australia (6):
  - Investigational Site Number : 0360007, St Leonards, New South Wales
  - Investigational Site Number :0360003, Woolloongabba, Queensland
  - Investigational Site Number :0360002, Kent Town, South Australia
  - Investigational Site Number :0360004, Hobart, Tasmania
  - Investigational Site Number :0360001, Fitzroy, Victoria
  - Investigational Site Number :0360006, Heidelberg West, Victoria
- Austria (4):
  - Investigational Site Number :0400003, Innsbruck
  - Investigational Site Number :0400001, Linz
  - Investigational Site Number :0400004, Linz
  - Investigational Site Number :0400002, Vienna
- Belarus (2):
  - Investigational Site Number :1120004, Vitebsk
  - Investigational Site Number :1120005, Vitebsk
- Belgium (8):
  - Investigational Site Number : 0560009, Brussels
  - Investigational Site Number :0560007, Brussels
  - Investigational Site Number :0560003, Edegem
  - Investigational Site Number : 0560004, Ghent
  - Investigational Site Number :0560006, Leuven
  - Investigational Site Number :0560008, Liège
  - Investigational Site Number :0560002, Mons
  - Investigational Site Number :0560001, Overpelt
- Bulgaria (7):
  - Investigational Site Number :1000002, Pleven
  - Investigational Site Number :1000005, Plovdiv
  - Investigational Site Number :1000004, Sofia
  - Investigational Site Number :1000008, Sofia
  - Investigational Site Number :1000001, Sofia
  - Investigational Site Number :1000006, Sofia
  - Investigational Site Number :1000009, Sofia
- Canada (11):
  - Investigational Site Number :1240017, Burnaby, British Columbia
  - Investigational Site Number :1240011, Halifax, Nova Scotia
  - Investigational Site Number :1240003, Ottawa, Ontario
  - Investigational Site Number :1240008, Toronto, Ontario
  - Investigational Site Number :1240006, Gatineau, Quebec
  - Investigational Site Number :1240005, Greenfield Park, Quebec
  - Investigational Site Number :1240004, Montreal, Quebec
  - Investigational Site Number :1240015, Montreal, Quebec
  - Investigational Site Number :1240007, Sherbrooke, Quebec
  - Investigational Site Number : 1240001, Québec
  - Investigational Site Number :1240021, Québec
- China (15):
  - Investigational Site Number :1560006, Beijing
  - Investigational Site Number :1560012, Beijing
  - Investigational Site Number :1560021, Beijing
  - Investigational Site Number :1560003, Beijing
  - Investigational Site Number :1560009, Beijing
  - Investigational Site Number :1560004, Changchun
  - Investigational Site Number :1560015, Changsha
  - Investigational Site Number :1560005, Chengdu
  - Investigational Site Number :1560019, Chongqing
  - Investigational Site Number :1560035, Fuzhou
  - Investigational Site Number :1560001, Guangzhou
  - Investigational Site Number :1560007, Hangzhou
  - Investigational Site Number :1560014, Shijiazhuang
  - Investigational Site Number :1560008, Taiyuan
  - Investigational Site Number :1560017, Xi'an
- Czechia (6):
  - Investigational Site Number :2030002, Brno
  - Investigational Site Number :2030004, Hradec Králové
  - Investigational Site Number :2030001, Jihlava
  - Investigational Site Number :2030010, Ostrava - Poruba
  - Investigational Site Number :2030005, Prague
  - Investigational Site Number :2030003, Teplice
- Denmark (3):
  - Investigational Site Number :2080001, Esbjerg
  - Investigational Site Number :2080005, Holstebro
  - Investigational Site Number :2080004, Odense
- Finland (3):
  - Investigational Site Number :2460003, Helsinki
  - Investigational Site Number :2460001, Tampere
  - Investigational Site Number :2460002, Turku
- France (14):
  - Investigational Site Number :2500011, Bron
  - Investigational Site Number :2500005, Clermont-Ferrand
  - Investigational Site Number :2500015, Gonesse
  - Investigational Site Number :2500009, Lille
  - Investigational Site Number :2500006, Montpellier
  - Investigational Site Number :2500008, Nancy
  - Investigational Site Number :2500010, Nantes
  - Investigational Site Number :2500017, Nîmes
  - Investigational Site Number :2500016, Paris
  - Investigational Site Number :2500014, Paris
  - Investigational Site Number :2500007, Paris
  - Investigational Site Number :2500003, Rennes
  - Investigational Site Number :2500001, Strasbourg
  - Investigational Site Number :2500012, Toulouse
- Germany (10):
  - Investigational Site Number :2760005, Bayreuth
  - Investigational Site Number :2760009, Berlin
  - Investigational Site Number :2760001, Dresden
  - Investigational Site Number :2760012, Essen
  - Investigational Site Number :2760002, Giessen
  - Investigational Site Number :2760010, Halle
  - Investigational Site Number :2760006, Hanover
  - Investigational Site Number :2760008, Münster
  - Investigational Site Number :2760004, Rostock
  - Investigational Site Number :2760011, Ulm
- Greece (7):
  - Investigational Site Number :3000001, Athens
  - Investigational Site Number :3000006, Athens
  - Investigational Site Number :3000002, Athens
  - Investigational Site Number :3000007, Athens
  - Investigational Site Number :3000004, Larissa
  - Investigational Site Number :3000003, Thessaloniki
  - Investigational Site Number :3000005, Thessaloniki
- Hungary (6):
  - Investigational Site Number :3480008, Budapest
  - Investigational Site Number :3480004, Budapest
  - Investigational Site Number :3480007, Budapest
  - Investigational Site Number :3480002, Pécs
  - Investigational Site Number :3480001, Szeged
  - Investigational Site Number :3480006, Tatabánya
- India (7):
  - Investigational Site Number :3560007, Gūrgaon
  - Investigational Site Number :3560003, Gūrgaon
  - Investigational Site Number :3560005, India
  - Investigational Site Number :3560004, Mangaluru
  - Investigational Site Number : 3560009, Nagpur
  - Investigational Site Number :3560006, New Delhi
  - Investigational Site Number :3560002, New Delhi
- Israel (5):
  - Investigational Site Number :3760002, Ashkelon
  - Investigational Site Number :3760003, Haifa
  - Investigational Site Number :3760008, Jerusalem
  - Investigational Site Number :3760004, Safed
  - Investigational Site Number :3760001, Tel Litwinsky
- Italy (12):
  - Investigational Site Number :3800011, Bergamo
  - Investigational Site Number :3800007, Cagliari
  - Investigational Site Number :3800012, Florence
  - Investigational Site Number :3800016, Florence
  - Investigational Site Number :3800014, Genova
  - Investigational Site Number :3800013, L’Aquila
  - Investigational Site Number :3800004, Milan
  - Investigational Site Number :3800001, Milan
  - Investigational Site Number :3800010, Milan
  - Investigational Site Number :3800008, Pavia
  - Investigational Site Number :3800005, Roma
  - Investigational Site Number :3800009, Roma
- Japan (12):
  - Investigational Site Number :3920016, Chiba, Chiba
  - Investigational Site Number :3920022, Morioka, Iwate
  - Investigational Site Number :3920011, Kyoto, Kyoto
  - Investigational Site Number :3920020, Sendai, Miyagi
  - Investigational Site Number :3920005, Niigata, Niigata
  - Investigational Site Number :3920004, Moriguchi-shi, Osaka
  - Investigational Site Number :3920001, Osaka, Osaka
  - Investigational Site Number :3920018, Kawagoe-shi, Saitama
  - Investigational Site Number :3920003, Kodaira-shi, Tokyo
  - Investigational Site Number :3920010, Ōta-ku, Tokyo
  - Investigational Site Number :3920009, Ube-shi, Yamaguchi
  - Investigational Site Number :3920023, Sagamihara-shi
- Lithuania (3):
  - Investigational Site Number :4400003, Kaunas
  - Investigational Site Number :4400002, Klaipėda
  - Investigational Site Number :4400001, Vilnius
- Netherlands (4):
  - Investigational Site Number :5280001, Amsterdam
  - Investigational Site Number :5280003, Breda
  - Investigational Site Number :5280006, Groningen
  - Investigational Site Number :5280002, Sittard-Geleen
- Norway (3):
  - Investigational Site Number :5780003, Bergen
  - Investigational Site Number :5780002, Namsos
  - Investigational Site Number :5780001, Oslo
- Poland (10):
  - Investigational Site Number :6160008, Plewiska, Greater Poland Voivodeship
  - Investigational Site Number :6160003, Bydgoszcz, Kuyavian-Pomeranian Voivodeship
  - Investigational Site Number :6160005, Warsaw, Masovian Voivodeship
  - Investigational Site Number :6160006, Warsaw, Masovian Voivodeship
  - Investigational Site Number :6160002, Katowice, Silesian Voivodeship
  - Investigational Site Number :6160007, Katowice, Silesian Voivodeship
  - Investigational Site Number :6160004, Katowice, Silesian Voivodeship
  - Investigational Site Number :6160001, Lodz
  - Investigational Site Number :6160012, Lublin
  - Investigational Site Number :6160011, Zabrze
- Portugal (6):
  - Investigational Site Number :6200001, Braga
  - Investigational Site Number :6200011, Lisbon
  - Investigational Site Number :6200007, Lisbon
  - Investigational Site Number :6200006, Lisbon
  - Investigational Site Number :6200002, Matosinhos Municipality
  - Investigational Site Number :6200010, Porto
- Romania (8):
  - Investigational Site Number :6420008, Bucharest
  - Investigational Site Number :6420004, Campulung Muscel
  - Investigational Site Number :6420006, Cluj-Napoca
  - Investigational Site Number :6420003, Constanța
  - Investigational Site Number :6420013, Oradea
  - Investigational Site Number :6420005, Sibiu
  - Investigational Site Number :6420001, Târgu Mureş
  - Investigational Site Number :6420002, Timișoara
- Russia (25):
  - Investigational Site Number :6430018, Barnaul
  - Investigational Site Number :6430025, Kaliningrad
  - Investigational Site Number :6430003, Kazan'
  - Investigational Site Number :6430022, Kemerovo
  - Investigational Site Number :6430017, Kirov
  - Investigational Site Number :6430024, Krasnoyarsk
  - Investigational Site Number :6430020, Moscow
  - Investigational Site Number :6430002, Moscow
  - Investigational Site Number :6430013, Moscow
  - Investigational Site Number :6430001, Moscow
  - Investigational Site Number :6430008, Moscow
  - Investigational Site Number :6430021, Nizhny Novgorod
  - Investigational Site Number :6430006, Nizhny Novgorod
  - Investigational Site Number :6430005, Novosibirsk
  - Investigational Site Number :6430026, Perm
  - Investigational Site Number :6430007, Pyatigorsk
  - Investigational Site Number :6430016, Rostov-on-Don
  - Investigational Site Number :6430011, Saint Petersburg
  - Investigational Site Number :6430004, Saint Petersburg
  - Investigational Site Number :6430009, Samara
  - Investigational Site Number :6430019, Saransk
  - Investigational Site Number :6430014, Smolensk
  - Investigational Site Number :6430012, Tyumen
  - Investigational Site Number :6430010, Ufa
  - Investigational Site Number :6430023, Yekaterinburg
- Spain (16):
  - Investigational Site Number :7240007, Seville, Andalusia
  - Investigational Site Number :7240013, Barcelona, Barcelona [Barcelona]
  - Investigational Site Number :7240016, Barcelona, Barcelona [Barcelona]
  - Investigational Site Number :7240012, Donostia / San Sebastian, Basque Country
  - Investigational Site Number :7240014, Salt, Girona [Gerona]
  - Investigational Site Number :7240017, Las Palmas de Gran Canaria, Las Palmas
  - Investigational Site Number :7240004, Majadahonda, Madrid
  - Investigational Site Number :7240001, Pozuelo de Alarcón, Madrid
  - Investigational Site Number :7240008, Córdoba
  - Investigational Site Number :7240015, Lleida
  - Investigational Site Number :7240005, Madrid
  - Investigational Site Number :7240002, Madrid
  - Investigational Site Number :7240003, Madrid
  - Investigational Site Number :7240009, Málaga
  - Investigational Site Number :7240010, Murcia
  - Investigational Site Number :7240011, Valencia
- Turkey (Türkiye) (12):
  - Investigational Site Number :7920005, Eskişehir
  - Investigational Site Number :7920010, Hatay
  - Investigational Site Number :7920002, Istanbul
  - Investigational Site Number :7920009, Istanbul
  - Investigational Site Number :7920007, Istanbul
  - Investigational Site Number :7920006, Istanbul
  - Investigational Site Number :7920003, Istanbul
  - Investigational Site Number :7920013, Izmir
  - Investigational Site Number :7920001, İzmit
  - Investigational Site Number :7920011, Kütahya
  - Investigational Site Number :7920012, Mersin
  - Investigational Site Number :7920008, Trabzon
- Ukraine (14):
  - Investigational Site Number :8040008, Chernivtsi
  - Investigational Site Number :8040016, Chernivtsi
  - Investigational Site Number :8040003, Dnipro
  - Investigational Site Number :8040010, Ivano-Frankivsk
  - Investigational Site Number :8040007, Kharkiv
  - Investigational Site Number :8040011, Kharkiv
  - Investigational Site Number :8040012, Kharkiv
  - Investigational Site Number :8040013, Kyiv
  - Investigational Site Number :8040005, Lutsk
  - Investigational Site Number :8040009, Lviv
  - Investigational Site Number :8040004, Lviv
  - Investigational Site Number :8040002, Odesa
  - Investigational Site Number :8040006, Vinnytsia
  - Investigational Site Number :8040014, Zhytomyr
- United Kingdom (11):
  - Investigational Site Number :8260003, Exeter, Devon
  - Investigational Site Number :8260008, Plymouth, Devon
  - Investigational Site Number :8260010, Swansea, Neath Port Talbot
  - Investigational Site Number :8260012, Nottingham, Nottinghamshire
  - Investigational Site Number :8260013, Oxford, Oxfordshire
  - Investigational Site Number :8260009, Bristol
  - Investigational Site Number :8260001, Cardiff
  - Investigational Site Number :8260005, London
  - Investigational Site Number :8260018, London
  - Investigational Site Number :8260014, Newcastle upon Tyne
  - Investigational Site Number :8260019, Salford

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- [Derived] Fox RJ, Bar-Or A, Traboulsee A, Oreja-Guevara C, Giovannoni G, Vermersch P, Syed S, Li Y, Vargas WS, Turner TJ, Wallstroem E, Reich DS; HERCULES Trial Group. Tolebrutinib in Nonrelapsing Secondary Progressive Multiple Sclerosis. N Engl J Med. 2025 May 15;392(19):1883-1892. doi: 10.1056/NEJMoa2415988. Epub 2025 Apr 8. PMID 40202696
- See also: EFC16645 Plain language Results Summary — https://sanofi.trialsummaries.com/Study/StudyDetails?id=25250&tenant=MT_SNY_9011

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 1438 participants were screened at 267 centers in 31 countries between 24-Sep-2020 and 02-Dec-2022, of which 307 were screen failures mainly due to not meeting eligibility criteria.
Pre-assignment Details: A total of 1131 participants were randomized in this study in a 2:1 ratio to receive either tolebrutinib or matching placebo in the double-blind (DB) period. Participants with 6-month confirmed disability progression (CDP) were given the option to receive open-label (OL) tolebrutinib. This was an event-driven (6-month CDP) trial with a variable treatment duration (end-of-study [EOS] duration: up to approximately 47 months).
Groups:
- DB: Placebo: Participants received placebo matched to tolebrutinib orally once daily up to approximately 47 months.
- DB: Tolebrutinib 60 mg: Participants received tolebrutinib 60 mg tablet orally once daily up to approximately 47 months.
- OL: Placebo/Tolebrutinib 60 mg: Participants who received placebo in DB period and achieved 6-month CDP were given the option to receive OL tolebrutinib 60 mg tablet orally once daily up to approximately 39 months in the OL.
- OL: Tolebrutinib 60 mg/Tolebrutinib 60 mg: Participants who received tolebrutinib 60 mg in DB period and achieved 6-month CDP were given the option to continue to receive OL tolebrutinib 60 mg tablet orally once daily up to approximately 39 months in the OL.
Period: DB Period
Arm/Group | DB: Placebo | DB: Tolebrutinib 60 mg | OL: Placebo/Tolebrutinib 60 mg | OL: Tolebrutinib 60 mg/Tolebrutinib 60 mg
Started (Randomized) | 377 | 754 | 0 | 0
Completed (Completed DB period) | 192 | 434 | 0 | 0
Not Completed | 185 | 320 | 0 | 0
Not completed — Other | 7 | 27 | 0 | 0
Not completed — Withdrawal by Subject | 67 | 122 | 0 | 0
Not completed — Progressive disease | 76 | 116 | 0 | 0
Not completed — Poor compliance to protocol | 1 | 5 | 0 | 0
Not completed — Lack of Efficacy | 19 | 19 | 0 | 0
Not completed — Adverse Event | 13 | 29 | 0 | 0
Not completed — Randomized and not treated | 2 | 2 | 0 | 0
Period: OL
Arm/Group | DB: Placebo | DB: Tolebrutinib 60 mg | OL: Placebo/Tolebrutinib 60 mg | OL: Tolebrutinib 60 mg/Tolebrutinib 60 mg
Started | 0 | 0 | 76 (Eligible participants switched to OL) | 120 (Eligible participants switched to OL)
Completed | 0 | 0 | 67 | 95
Not Completed | 0 | 0 | 9 | 25
Not completed — Withdrawal by Subject | 0 | 0 | 6 | 17
Not completed — Progressive disease | 0 | 0 | 1 | 2
Not completed — Poor compliance to protocol | 0 | 0 | 1 | 0
Not completed — Adverse Event | 0 | 0 | 1 | 0
Not completed — Other | 0 | 0 | 0 | 6

BASELINE CHARACTERISTICS:
Population: Analysis was performed on randomized population.
Groups:
- Total: Total of all reporting groups
Arm/Group | DB: Placebo | DB: Tolebrutinib 60 mg | Total
Number analyzed (Participants) | 377 | 754 | 1131
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.9 (8.0) | 48.9 (8.0) | 48.9 (8.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 242 | 454 | 696
  Male | 135 | 300 | 435
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 19 | 36 | 55
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 6 | 10
  White | 348 | 703 | 1051
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 6 | 7 | 13

OUTCOME MEASURES:

1. Primary Outcome: Time to Onset of 6-Month Confirmed Disability Progression (CDP) as Assessed by Expanded Disability Status Scale (EDSS)
Description: The EDSS is a disability scale that assesses the following 7 functional domains: visual, brainstem, pyramidal [motor], cerebellar [coordination], sensory, cerebral, and bowel/bladder. The total EDSS ranges from 0 (normal) to 10 (death due to multiple sclerosis [MS]) (0.5 increments from 1-10; next increase after 0 is 1). Higher scores indicated increased disability. Time to onset of 6-month CDP was defined as the time from randomization to the onset of a sustained increase from baseline in EDSS score of >=1.0 point from the baseline EDSS score when the baseline score was <=5.0 or of >=0.5 points when the baseline EDSS score was >5.0 confirmed after a minimum 6-month interval.
Time Frame: Baseline (Day 1) up to approximately 47 months
Population: The intent-to-treat (ITT) population included all randomized participants according to the intervention group allocated by the randomization, irrespective of the study intervention received.
Measure: Median (Full Range); unit: months
Arm/Group | DB: Placebo | DB: Tolebrutinib 60 mg
Number analyzed (Participants) | 377 | 754
months | 11.97 [0.5 to 39.1] | 12.04 [2.8 to 37.4]
Statistical Analysis 1: Comparison: DB: Placebo vs DB: Tolebrutinib 60 mg; Derived using Cox proportional-hazards model with robust variance estimation.Covariates were treatment group,age at screening (>40,<=40 years),geographic region (United States [US], non-US),baseline EDSS score & baseline gadolinium (Gd)-enhancing T1 lesions (presence, absence).In this analysis, for participants who completed study with 3-month confirmation and continued to meet disability progression criteria throughout EOS, their 6-month CDP status was imputed via multiple imputation method; Test type: Superiority — A hierarchical testing procedure was used to control the overall type I error. Testing was then performed sequentially in order the outcome measures are reported and continued when previous outcome measure was statistically significant at 2-sided 0.05. Primary and first 6 secondary endpoints are included in this procedure; p = 0.0026, Regression, Cox — Threshold for significance at 2-sided 0.05 level; Hazard Ratio (HR) = 0.693, 95% CI 2-sided [0.546 to 0.880]

2. Secondary Outcome: Time to Onset of 3-month Confirmed Disability Progression as Assessed by Expanded Disability Status Scale
Description: The EDSS is a disability scale that assesses the following 7 functional domains: visual, brainstem, pyramidal [motor], cerebellar [coordination], sensory, cerebral, and bowel/bladder. The total EDSS ranges from 0 (normal) to 10 (death due to MS) (0.5 increments from 1-10; next increase after 0 is 1). Higher scores indicated increased disability. Time to onset of 3-month CDP was defined as the time from randomization to the onset of a sustained increase from baseline in EDSS score (of >=1.0 point from the baseline EDSS score when the baseline score is <=5.0, of >=0.5 points when the baseline EDSS score is >5.0) confirmed after a minimum 3-month interval. The confirmation of 3-month CDP followed the same criteria as that of 6-month CDP.
Time Frame: Baseline (Day 1) up to approximately 47 months
Population: The ITT population included all randomized participants according to the intervention group allocated by the randomization, irrespective of the study intervention received.
Measure: Median (Full Range); unit: months
Arm/Group | DB: Placebo | DB: Tolebrutinib 60 mg
Number analyzed (Participants) | 377 | 754
months | 11.96 [0.5 to 39.1] | 12.04 [2.8 to 39.5]
Statistical Analysis 1: Comparison: DB: Placebo vs DB: Tolebrutinib 60 mg; Derived using Cox proportional-hazards model with robust variance estimation. Covariates were treatment group, age at screening (>40, <=40 years), geographic region (US, non-US), baseline EDSS score and baseline Gd-enhancing T1 lesions (presence, absence); Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.0134, Regression, Cox — Threshold for significance at 2-sided 0.05 level; Hazard Ratio (HR) = 0.757, 95% CI 2-sided [0.607 to 0.944]

3. Secondary Outcome: Mean Number of New and/or Enlarging T2-hyperintense Lesions Per Year
Description: Magnetic resonance imaging (MRI) of the brain was performed to identify number of new and/or enlarging T2-hyperintense lesions defined as the sum of the individual number of new and/or enlarging T2 lesions from baseline up to and including the EOS visit.
Time Frame: Baseline (Day 1) up to approximately 47 months
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: number of T2 lesions
Arm/Group | DB: Placebo | DB: Tolebrutinib 60 mg
Number analyzed (Participants) | 377 | 754
number of T2 lesions | 2.948 [2.239 to 3.880] | 1.835 [1.441 to 2.336]
Statistical Analysis 1: Comparison: DB: Placebo vs DB: Tolebrutinib 60 mg; Derived using negative binomial model with the number of new and/or enlarging T2-hyperintense lesions between randomization date and EOS date as the response variable, treatment group, age at screening (>40, <=40 years), geographic region (US, non-US), baseline EDSS score, and baseline number of T2 lesions as covariates, and log transformed observation duration as the offset variable; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.0110, Chi-squared — Threshold for significance at 2-sided 0.05 level; Relative Risk = 0.622, 95% CI 2-sided [0.432 to 0.897]

4. Secondary Outcome: Time to Onset of Sustained 20% Increase in the 9-hole Peg Test (HPT) for at Least 3 Months
Description: The 9-HPT is a brief, standardized, quantitative test of upper extremity function and the time to complete the 9-HPT is used to assess a participant's manual dexterity and fine motor skills. A participant was asked to place the pegs into the holes and remove them with the dominant and non-dominant hand; two successful trials for each hand. The amount of time (in seconds) required to place and remove all nine pegs was recorded for each trial (ranging from 10 to 300 seconds). The mean time to test completion served for assessment of the participant's hand dexterity. Higher value indicated worse outcome. An increase of >20% from the baseline in the 9-HPT was considered meaningful worsening; time to onset of sustained 20% increase for at least 3 months is presented.
Time Frame: Baseline (Day 1) up to approximately 47 months
Population: as for outcome 2
Measure: Median (Full Range); unit: months
Arm/Group | DB: Placebo | DB: Tolebrutinib 60 mg
Number analyzed (Participants) | 377 | 754
months | 12.39 [2.5 to 33.3] | 12.21 [2.8 to 39.2]
Statistical Analysis 1: Comparison: DB: Placebo vs DB: Tolebrutinib 60 mg; [analysis description as in outcome 2, analysis 1]; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.8428, Regression, Cox — Threshold for significance at 2-sided 0.05 level; Hazard Ratio (HR) = 0.972, 95% CI 2-sided [0.735 to 1.286]

5. Secondary Outcome: Time to Onset of Sustained 20% Increase in the Timed 25-foot Walk (T25-FW) for at Least 3 Months
Description: The T25-FW test is a quantitative mobility and leg function performance test used to assess a participant's walking ability. A participant was directed to one end of a clearly marked 25-foot course and instructed to walk 25 feet as quickly as safely possible for 2 trials. The amount of time (in seconds) to walk 25 feet was recorded (ranging from 2.2 to 180 seconds). The mean walk time was used for assessment of the participant's walking ability. Higher value indicated worse outcome. An increase of >20% from the baseline in the T25-FW test was considered meaningful worsening; time to onset of sustained 20% increase for at least 3 months is presented.
Time Frame: Baseline (Day 1) up to approximately 47 months
Population: as for outcome 2
Measure: Median (Full Range); unit: months
Arm/Group | DB: Placebo | DB: Tolebrutinib 60 mg
Number analyzed (Participants) | 377 | 754
months | 9.25 [2.5 to 36.3] | 9.54 [2.8 to 39.3]
Statistical Analysis 1: Comparison: DB: Placebo vs DB: Tolebrutinib 60 mg; [analysis description as in outcome 2, analysis 1]; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.0040, Regression, Cox; Hazard Ratio (HR) = 0.767, 95% CI 2-sided [0.640 to 0.919]

6. Secondary Outcome: Time to Onset of 6-month Confirmed Disability Improvement (CDI) as Assessed by Expanded Disability Status Scale
Description: The EDSS is a disability scale that assesses the following 7 functional domains: visual, brainstem, pyramidal [motor], cerebellar [coordination], sensory, cerebral, and bowel/bladder. The total EDSS ranges from 0 (normal) to 10 (death due to MS) (0.5 increments from 1-10; next increase after 0 is 1). Higher scores indicated increased disability. CDI was defined as a >=1 point decrease in the EDSS score from baseline confirmed over at least 6 months.
Time Frame: Baseline (Day 1) up to approximately 47 months
Population: as for outcome 2
Measure: Median (Full Range); unit: months
Arm/Group | DB: Placebo | DB: Tolebrutinib 60 mg
Number analyzed (Participants) | 377 | 754
months | 12.04 [3.0 to 24.1] | 11.89 [2.9 to 33.0]
Statistical Analysis 1: Comparison: DB: Placebo vs DB: Tolebrutinib 60 mg; [analysis description as in outcome 2, analysis 1]; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.0206, Regression, Cox; Hazard Ratio (HR) = 1.882, 95% CI 2-sided [1.102 to 3.214]

7. Secondary Outcome: Percent Change in Brain Volume at EOS Compared to Month 6
Description: MRI of the brain was performed to evaluate percent change in brain volume which is considered as a marker of the central nervous system degenerative process. Least squares (LS) mean is presented.
Time Frame: Month 6 to EOS (up to approximately 47 months)
Population: The ITT population included all randomized participants according to the intervention group allocated by the randomization, irrespective of the study intervention received. Only those participants with data collected at specified timepoints are reported.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | DB: Placebo | DB: Tolebrutinib 60 mg
Number analyzed (Participants) | 223 | 451
percent change | -0.776 (0.0479) | -0.694 (0.0336)
Statistical Analysis 1: Comparison: DB: Placebo vs DB: Tolebrutinib 60 mg; Covariates in the mixed-effect model with repeated measures were treatment group, age at screening (>40, <=40 years), geographic region (US, non-US), visit, treatment-by-visit interaction, cube root transformed Month 6 brain volume, and cube root transformed Month 6 brain volume-by-visit interaction; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.1646, Mixed model repeated measures (MMRM); LS Mean Difference = 0.082, 95% CI 2-sided [-0.034 to 0.197]

8. Secondary Outcome: Change From Baseline in Cognitive Function as Assessed by Symbol Digit Modalities Test (SDMT) at EOS
Description: The SDMT is used to assess processing speed, divided attention, visual scanning, tracking and motor speed. It involves a simple substitution task using a reference key. The number of correct substitutions and number of items completed within a 90 second interval (maximum 110 seconds) are recorded. A decrease of 4 points from baseline on the SDMT is considered meaningful worsening. The score was the number of correctly coded items from 0-110 in 90 seconds; higher scores indicated better outcome. LS mean is presented. Baseline was defined as the last available value prior to the first dose of study intervention.
Time Frame: Baseline (Day 1) to EOS (up to approximately 47 months)
Population: as for outcome 7
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | DB: Placebo | DB: Tolebrutinib 60 mg
Number analyzed (Participants) | 271 | 546
score on a scale | 0.171 (0.0373) | 0.136 (0.0264)

9. Secondary Outcome: Change From Baseline in Cognitive Function as Assessed by California Verbal Learning Test Second Edition (CVLT-II) at EOS
Description: The CVLT-II is a verbal learning and memory test consisting of recall and recognition of a list of 16 words. The list was read by the examiner, participants listened to the list and reported as many of the items as possible. For each assessment, 5 trials were completed. Standardized scores were used for analysis. The maximum possible score was 80 and a minimum was 0. A higher score indicated better recall meaning improved cognitive function. LS mean is presented. Baseline was defined as the last available value prior to the first dose of study intervention.
Time Frame: Baseline (Day 1) to EOS (up to approximately 47 months)
Population: as for outcome 7
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | DB: Placebo | DB: Tolebrutinib 60 mg
Number analyzed (Participants) | 262 | 531
score on a scale | 13.448 (0.9571) | 14.169 (0.6759)

10. Secondary Outcome: Change From Baseline in Multiple Sclerosis Quality of Life-54 (MSQoL-54) Questionnaire Score at EOS
Description: MSQoL-54 is standardized instrument with generic and MS-specific items which generates 12 subscales & 2 single-item measures (satisfaction with sexual function [1 item] & change in health [1 item].12 subscales are as follows:a:physical health (10 items),b:health perceptions (5 items), c:energy (5 items),d:role limitation physical (4 items),e:sexual function (4 items),f:pain (3 items),g:social function (3 items),h:health distress (4 items),i:overall quality of life (2 items),j:emotional well-being (5 items),k:role limitations emotional (3 items) and l:cognitive function (4 items).Physical health composite score was calculated as weighted sum of 'a to h' subscales and mental health composite score was calculated as weighted sum of 'i to l' subscales mentioned above.Each composite score was transformed linearly to common 0 (worst) to 100 (best) score range;LS mean is presented.Higher score indicated improved QoL.Baseline:last available value prior to first dose of study intervention.
Time Frame: Baseline (Day 1) to EOS (up to approximately 47 months)
Population: as for outcome 7
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | DB: Placebo | DB: Tolebrutinib 60 mg
Number analyzed (Participants) | 268 | 552
score on a scale
  Physical health composite score: number analyzed (Participants) | 262 | 536
  Physical health composite score | -3.979 (0.8032) | -3.455 (0.5623)
  Mental health composite score | -4.648 (0.9964) | -3.944 (0.6959)

11. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (AEs), Treatment-emergent Serious AEs, Treatment-emergent AEs Leading to Permanent Study Intervention Discontinuation, and Treatment-emergent Adverse Events of Special Interest (AESIs)
Description: An AE was any untoward medical occurrence in a participant or clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. SAE was any untoward medical occurrence that at any dose: resulted in death, was life-threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent disability/incapacity, was a congenital anomaly/birth defect or was an important medical event. An AESI was an AE (serious or nonserious) of scientific and medical concern specific to the Sponsor's product or program for which ongoing monitoring and immediate notification by the Investigator to the Sponsor was required. TEAEs were defined as AEs that developed, worsened or became serious during the TE period.
Time Frame: From first dose of study intervention (Day 1) up to end of follow-up, up to approximately 47 months
Population: The safety population included all randomized participants exposed to study intervention, regardless of the amount of exposure, analyzed according to the intervention actually received.
Measure: Count of Participants; unit: Participants
Arm/Group | DB: Placebo | DB: Tolebrutinib 60 mg | OL: Placebo/Tolebrutinib 60 mg | OL: Tolebrutinib 60 mg/Tolebrutinib 60 mg
Number analyzed (Participants) | 375 | 752 | 76 | 120
Participants
  TEAEs | 293 | 613 | 47 | 80
  TESAEs | 39 | 113 | 9 | 11
  TEAEs Leading to Permanent Study Intervention Discontinuation | 11 | 29 | 1 | 0
  TEAESIs | 20 | 75 | 6 | 10

12. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of Tolebrutinib and M2 Metabolite
Description: Blood samples were collected at specified timepoints to assess Cmax of tolebrutinib and M2 metabolite using a population pharmacokinetics (PopPK) model.
Time Frame: 30-90 minutes post-dose at Months 6, 9, and 12 and 2.5-5 hours post-dose at Months 6 and 12
Population: The PK population included all participants in the safety population with at least 1 non-missing PK sample after first dose of the study intervention. Only those participants with data collected at specified timepoints are reported.
Measure: Mean (Standard Deviation); unit: nanogram/milliliter (ng/mL)
Arm/Group | DB: Tolebrutinib 60 mg
Number analyzed (Participants) | 669
nanogram/milliliter (ng/mL)
  Tolebrutinib | 9.94 (6.18)
  M2 Metabolite | 27.5 (17.3)

13. Secondary Outcome: Time to Maximum Observed Plasma Concentration (Tmax) of Tolebrutinib and M2 Metabolite
Description: Blood samples were collected at specified timepoints to assess Tmax of tolebrutinib and M2 metabolite using a PopPK model.
Time Frame: 30-90 minutes post-dose at Months 6, 9, and 12 and 2.5-5 hours post-dose at Months 6 and 12
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: hour (h)
Arm/Group | DB: Tolebrutinib 60 mg
Number analyzed (Participants) | 669
hour (h)
  Tolebrutinib | 1.42 (0.674)
  M2 Metabolite | 1.52 (0.667)

14. Secondary Outcome: Area Under the Plasma Concentration-time Curve Over the Last 24-hours Dosing Interval (AUC0-24) of Tolebrutinib and M2 Metabolite
Description: Blood samples were collected at specified timepoints to assess AUC0-24 of tolebrutinib and M2 metabolite using a PopPK model.
Time Frame: 30-90 minutes post-dose at Months 6, 9, and 12 and 2.5-5 hours post-dose at Months 6 and 12
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | DB: Tolebrutinib 60 mg
Number analyzed (Participants) | 669
ng*h/mL
  Tolebrutinib | 29.6 (17.8)
  M2 Metabolite | 84.6 (53.7)

15. Secondary Outcome: Change From Baseline in Plasma Neurofilament Light Chain (NfL) and Serum Chitinase-3 Like Protein-1 (Chi3L1) Levels at EOS
Description: Blood samples were collected at specified timepoints to assess change from baseline in NfL and Chi3L1. Baseline was defined as the last available value prior to the first dose of study intervention.
Time Frame: Baseline (Day 1) to EOS (up to approximately 47 months)
Population: The safety population included all randomized participants exposed to study intervention, regardless of the amount of exposure, analyzed according to the intervention actually received. Only those participants with data collected at specified timepoints are reported.
Measure: Median (Inter-Quartile Range); unit: picogram/mL
Arm/Group | DB: Placebo | DB: Tolebrutinib 60 mg
Number analyzed (Participants) | 171 | 410
picogram/mL
  NfL: number analyzed (Participants) | 168 | 403
  NfL | 1.070 [-1.285 to 3.615] | 1.900 [-0.370 to 4.470]
  Chi3L1 | 5156.900 [-1555.700 to 12099.200] | 3132.250 [-2822.100 to 13407.100]

16. Secondary Outcome: Change From Baseline in Cluster of Differentiation (CD)19+ B Cells at EOS
Description: Blood samples were collected at specified timepoints to assess change from baseline in CD19+ B cells. Baseline was defined as the last available value prior to the first dose of study intervention.
Time Frame: Baseline (Day 1) to EOS (up to approximately 47 months)
Population: as for outcome 15
Measure: Median (Inter-Quartile Range); unit: cells/microliter
Arm/Group | DB: Placebo | DB: Tolebrutinib 60 mg
Number analyzed (Participants) | 26 | 58
cells/microliter | 10.000 [-18.000 to 77.000] | -63.000 [-105.000 to -8.000]

17. Secondary Outcome: Change From Baseline in Serum Immunoglobulin (Ig) Levels at EOS
Description: Blood samples were collected at specified timepoints to assess change from baseline in IgG and IgM levels. Baseline was defined as the last available value prior to the first dose of study intervention.
Time Frame: Baseline (Day 1) to EOS (up to approximately 47 months)
Population: as for outcome 15
Measure: Median (Inter-Quartile Range); unit: gram/liter
Arm/Group | DB: Placebo | DB: Tolebrutinib 60 mg
Number analyzed (Participants) | 149 | 323
gram/liter
  IgG: number analyzed (Participants) | 149 | 320
  IgG | 0.350 [-0.280 to 1.310] | -0.085 [-0.845 to 0.665]
  IgM: number analyzed (Participants) | 142 | 323
  IgM | 0.050 [-0.080 to 0.150] | -0.240 [-0.450 to -0.120]

ADVERSE EVENTS:
Time Frame: From first dose of study intervention (Day 1) up to end of follow-up, up to approximately 47 months
Description: Analysis was performed on safety population. All-cause mortality was performed on randomized population. This was an event-driven (6-month CDP) trial with a variable treatment duration, EOS: up to approximately 47 months.
Arm/Group | DB: Placebo | DB: Tolebrutinib 60 mg | OL: Placebo/Tolebrutinib 60 mg | OL: Tolebrutinib 60 mg/Tolebrutinib 60 mg
All-Cause Mortality (participants affected / at risk) | 1/377 | 2/754 | 0/76 | 0/120
Serious Adverse Events (participants affected / at risk) | 39/375 | 113/752 | 9/76 | 11/120
Other Adverse Events (participants affected / at risk) | 182/375 | 368/752 | 25/76 | 41/120
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DB: Placebo (N=375) | DB: Tolebrutinib 60 mg (N=752) | OL: Placebo/Tolebrutinib 60 mg (N=76) | OL: Tolebrutinib 60 mg/Tolebrutinib 60 mg (N=120)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Bacterial Pyelonephritis (Infections and infestations) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Covid-19 (Infections and infestations) | 0 (0) | 7 (7) | 1 (1) | 1 (1)
Covid-19 Pneumonia (Infections and infestations) | 2 (2) | 8 (8) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cystitis (Infections and infestations) | 1 (1) | 2 (3) | 0 (0) | 0 (0)
Cystitis Bacterial (Infections and infestations) | 2 (2) | 1 (3) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis Viral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Herpes Zoster (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 3 (3) | 5 (5) | 0 (0) | 1 (1)
Pneumonia Bacterial (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Pneumonia Pneumococcal (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia Viral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyelonephritis (Infections and infestations) | 0 (0) | 3 (3) | 1 (1) | 0 (0)
Pyelonephritis Acute (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pyelonephritis Chronic (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory Tract Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Upper Respiratory Tract Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Upper Respiratory Tract Infection Bacterial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 1 (3) | 3 (3) | 0 (0) | 2 (2)
Urosepsis (Infections and infestations) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Varicella Zoster Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Viral Upper Respiratory Tract Infection (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Wound Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Benign Neoplasm Of Thyroid Gland (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bladder Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bladder Cancer Stage 0, With Cancer In Situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Chronic Myeloid Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Endometrial Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lung Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Prostate Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Renal Cell Carcinoma Stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Squamous Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Uterine Leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Delirium (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Suicide Attempt (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Brain Hypoxia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Brain Oedema (Nervous system disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Generalised Tonic-Clonic Seizure (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intracranial Hypotension (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ischaemic Stroke (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Loss Of Consciousness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lumbar Radiculopathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Monoparesis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Multiple Sclerosis (Nervous system disorders) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
Multiple Sclerosis Pseudo Relapse (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Multiple Sclerosis Relapse (Nervous system disorders) | 0 (0) | 8 (8) | 0 (0) | 0 (0)
Muscle Spasticity (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Optic Neuritis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Parkinsonian Gait (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Post-Traumatic Headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Restless Legs Syndrome (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Sciatica (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Secondary Progressive Multiple Sclerosis (Nervous system disorders) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Subarachnoid Haemorrhage (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Trigeminal Neuralgia (Nervous system disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Vertigo Cns Origin (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Retinal Detachment (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Uveitis (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Visual Field Defect (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute Vestibular Syndrome (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vertigo Positional (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute Myocardial Infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Atrial Fibrillation (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Left Ventricular Dysfunction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myocardial Infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sinus Node Dysfunction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumothorax Spontaneous (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal Pain Lower (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Duodenal Ulcer Haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Faecaloma (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Functional Gastrointestinal Disorder (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastric Ulcer Haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haematemesis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haemorrhoidal Haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Megacolon (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Obstructive Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Terminal Ileitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Upper Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cholecystitis Acute (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Drug-Induced Liver Injury (Hepatobiliary disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Gallbladder Polyp (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hepatic Failure (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chondropathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (3) | 0 (0) | 1 (1)
Neck Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute Kidney Injury (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Renal Colic (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acquired Hydrocele (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Benign Prostatic Hyperplasia (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cervical Dysplasia (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gait Disturbance (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Malaise (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oedema Peripheral (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rebound Effect (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Alanine Aminotransferase Increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiac Murmur (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ankle Fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Brain Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cervical Vertebral Fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Craniocerebral Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Extradural Haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (2) | 3 (3) | 0 (0) | 1 (1)
Femoral Neck Fracture (Injury, poisoning and procedural complications) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Femur Fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Fibula Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hip Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Humerus Fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Intentional Overdose (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Joint Dislocation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Limb Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lumbar Vertebral Fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Pelvic Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Post-Traumatic Pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Radius Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rib Fracture (Injury, poisoning and procedural complications) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Road Traffic Accident (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Shoulder Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin Laceration (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skull Fractured Base (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Spinal Compression Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Subcutaneous Haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tibia Fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Traumatic Haemothorax (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Traumatic Liver Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ulna Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Assisted Suicide (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rehabilitation Therapy (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DB: Placebo (N=375) | DB: Tolebrutinib 60 mg (N=752) | OL: Placebo/Tolebrutinib 60 mg (N=76) | OL: Tolebrutinib 60 mg/Tolebrutinib 60 mg (N=120)
Covid-19 (Infections and infestations) | 85 (96) | 185 (225) | 4 (4) | 14 (14)
Influenza (Infections and infestations) | 13 (14) | 41 (60) | 2 (2) | 5 (6)
Nasopharyngitis (Infections and infestations) | 26 (35) | 70 (94) | 2 (3) | 8 (10)
Urinary Tract Infection (Infections and infestations) | 49 (81) | 82 (152) | 14 (22) | 12 (19)
Headache (Nervous system disorders) | 27 (31) | 54 (79) | 2 (2) | 4 (4)
Arthralgia (Musculoskeletal and connective tissue disorders) | 19 (21) | 49 (55) | 0 (0) | 2 (2)
Back Pain (Musculoskeletal and connective tissue disorders) | 24 (25) | 47 (56) | 1 (1) | 3 (3)
Accidental Overdose (Injury, poisoning and procedural complications) | 19 (22) | 25 (29) | 0 (0) | 3 (3)
Fall (Injury, poisoning and procedural complications) | 40 (54) | 70 (106) | 4 (4) | 6 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor supports publication of clinical trial results but may request that investigators temporarily delay or alter publications in order to protect proprietary information. The Sponsor may also require that the results of multicenter studies be published only in their entirety and not as individual site data.

DOCUMENTS (2):
  • Study Protocol (2023-12-20): https://cdn.clinicaltrials.gov/large-docs/41/NCT04411641/Prot_000.pdf
  • Statistical Analysis Plan (2024-04-30): https://cdn.clinicaltrials.gov/large-docs/41/NCT04411641/SAP_001.pdf